#### AMC PROTOCOL #084 MODEL INFORMED CONSENT FORM

Study Title for Study Participants: Testing methods to screen HIV-positive women for

predictors of anal cancer

Official Study Title for Internet

Search on http://www.ClinicalTrials.gov: Screening HIV Infected Women for Anal Cancer

**Precursors** 

## A Multi-Center Trial of the AIDS Malignancy Clinical Trials Consortium (AMC)

Cancer of the cervix (cervical cancer) and cancer of the anus (anal cancer) are caused by the human papillomavirus, or HPV. HPV is a virus that can infect and grow within the cervix, anus, vagina, and vulva. HPV infections are very common in HIV-positive women. Sometimes HPV can cause changes in some of the cells. When this happens in the cervix or the anus, the areas of changed cells are called high-grade intraepithelial lesions, or HSIL. Cervical and anal HSIL will sometimes turn into cancer. Treating HSIL helps to prevent cancer. People with HIV infection have a higher risk of getting HSIL and cancer.

## What is the usual approach to screen HIV-positive women for predictors for anal cancer?

You are being asked to take part in this study because you are an adult woman and you are infected with HIV. Women with HIV are at higher risk for getting a cancer related to human papillomavirus (HPV) compared with women who don't have HIV. There is no standard for screening for anal HSIL or cancer. Methods to screen women for HSIL or anal cancer vary at different centers. They may include rectal exams, doing a Pap (cytology) test of the anus, or waiting to see if any HSIL lesions get worse.

## What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example, you may seek care (cervical / anal Pap test, etc.) from your primary care provider. You may choose to have no screening for anal HSIL or cancer.

Your doctor may be part of this study team. As part of the study team, your doctor is interested in your clinical welfare and also the study. You may ask for a second opinion about your care from another doctor at any time before or during the study. You do not have to take part in any research study offered by your doctor.

#### Why is this study being done?

The purpose of this study is to figure out the best screening test to find HPV and HSIL cell changes in the anus in HIV-positive women. We want to know if the anal Pap test by itself or the anal Pap test along with anal HPV tests is better at finding cell changes in the anus. This study was designed to find out whether an anal Pap (cytology) will help HIV-positive women. The

study will also help to figure out what may put you at higher risk for anal HSIL. The overall goal of the study is to find the best way to screen for anal cancer in HIV-positive women.

# What are the study groups?

This is a cohort study. In cohort studies, researchers follow participants over time to observe changes in their health. All study participants will have the same tests and procedures. It will include study visits for anal exams and screening tests every 6 months for up to 2 years.

You will be one of approximately [insert local accrual estimate] subjects to be asked to participate at this location. The study will take place at up to 14 centers across the U.S. A total of 300 HIV-positive women will take part in this study at all sites.

## How long will I be in this study?

If you agree to take part, you may be in the study for up to 2 years. After your first study visit, you will be asked to come back every 6 months, for a total of 5 study visits. However, if you have HSIL (changed cells in your anus) at any visit, you will be referred for treatment and will no longer be part of the study.

## What extra tests and procedures will I have if I take part in this study?

If you agree to take part and sign the consent form, the research staff will review your medical records to find out if you qualify. If you qualify, you will have the tests and evaluations listed below.

- We will ask questions about your medical history, HIV symptoms, medications, and any allergies. Tell the doctor if you have an allergy to lidocaine.
- You will have a urine pregnancy test if you are able to become pregnant.
- The study doctor will do an anal and genital exam. During the exam you will have a cervical Pap and HPV tests (similar to tests you have for routine medical care), anal Pap and HPV tests
  - Ouring the anal Pap, the study doctor will collect anal cells with three swabs. The swab looks like a Q-tip. Each swab is soaked in water and placed an inch or two into the anus, one at a time. The clinician will slowly remove the swab and turn it in a spiral motion with mild pressure on the anal wall. The clinician will place each of the swabs into a small bottle with fluid to preserve the cells. Doctors will then look at the anal cells under a microscope to look for HSIL and anal cancer. We will also test the samples for HPV in different ways.
- An exam called High Resolution Anoscopy, or HRA, and anal biopsies
  - During the HRA, the study doctor will insert a lubricated plastic anoscope to look into the anus for abnormal areas. The provider will apply a swab dipped in acetic acid (dilute vinegar) and/or iodine to the skin inside the anus to help see any abnormal areas. The study doctor will use a colposcope (a machine with a magnifying lens) to see the skin inside the anus.
  - O During the anal biopsy, the study doctor will take at least 2 small pieces of anal tissue (the size of a sesame seed). The study doctor may give you a lidocaine injection to numb

the tissue before taking the biopsy. Please tell the study doctor if you are allergic to seafood, shellfish, contrast dye for a CAT scan, iodine, lidocaine, novocaine, or tetracaine. The study doctor will take the biopsy from any areas that are worrisome for HSIL and anal cancer. If no areas look abnormal, the study doctor will take 2 biopsies from different areas to rule out HSIL or anal cancer. We will send the tissue to a laboratory to look for HSIL and anal cancer.

- You will also have some blood (1 tablespoon) drawn for tests that measure how your HIV is affecting your health.
- We will ask you if you would like to donate blood to the AIDS and Cancer Specimen Resource (ACSR). If you agree, you will sign another consent form. If you don't agree, it will not prevent you from taking part in this study.
- We will give you a questionnaire about your smoking status, sexual history, medical history, and how the study procedures (anal Pap and HRA) make you feel.

You will be asked to return every six months for 2 years follow-up visits. During each visit we will ask you to fill out a questionnaire and you will have a repeat anal Pap and anal HPV testing. At visits 3 (1 year) and 5 (2 years), you will also have a repeat cervical Pap, cervical HPV test, blood tests, and high-resolution anoscopy. After every study visit, we will call you within two weeks after the visit and ask you questions about the study procedures and how they made you feel and any side effects you may have had from them.

If you have an abnormal anal biopsy tests, then we will recommend follow-up care for you. You can stay in the study and your study visits will continue unless you have HSIL (areas of changed cells) because you would need to be treated by your doctor. If you have an abnormal cervical Pap, we will recommend follow-up care while you continue in the study.

Each study visit may take up to 2 hours. Extra time may be needed for extra visits if the doctor or nurse feels these are important for your health. The time needed to participate in this study is 10 hours total for the 2 year study period.

#### Will you get the results of the tests done on your specimens?

We will give you and your doctor the results of your cervical and anal Pap tests, and biopsies. We will call you on the phone with the results in about 4 weeks. If you are not reachable by phone, then we will mail the results to you.

The doctor or nurse will advise you if there are any further steps to take and will schedule any follow-up appointments needed. Any follow-up appointments for abnormal results are considered standard of care and not related to this research study. If you have abnormal results, you will need to discuss the results with your doctor.

We will send some of your specimens to labs at three companies outside of this medical center. These labs are at Gen-Probe, Inc., QIAGEN Sciences, LLC, and Arbor Vita Corporation. They will run three different kinds of tests for HPV. They may also test samples for other biomarkers (biologic substances) related to HPV infection. Your samples will be identified with code numbers and kept completely private.

We will not give you the results of HPV testing during the study. This is because the tests are experimental and the meaning of HPV test results for your medical care is not known. We will tell you if there is any new information for this study that may affect your health, welfare, or your decision to stay in this study.

## What possible risks can I expect from taking part in this study?

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. You should tell your study doctor about any side effects that you have while taking part in the study.

Risks of questionnaires: There is a chance that you may feel embarrassed or uneasy by the personal nature of the questions asked in the study. If so, let the researcher know.

Risks of anal Pap test: There may be discomfort, pressure, and/or urgency to have a bowel movement during the procedure, and occasional bleeding.

Risks related to high resolution anoscopy and anal biopsy:

- Placing the anoscope may cause mild discomfort
- Applying acetic acid (dilute vinegar) and iodine to the anal tissue may cause minor discomfort
- Injecting lidocaine or other pain medicine to take a biopsy may cause minor discomfort. Lidocaine risks include a pinching or burning sensation from the injection. There is a very slight incidence of reaction to the anesthetic including rash, flushing, rapid heartbeat and dizziness.
- Taking an anal biopsy may cause temporary discomfort. There is a very slight risk of infection from the anal biopsy (less than 1%). Contact the study clinic if you have symptoms of infection (fever, redness, or swelling).
- Minor bleeding can happen after each biopsy. We will stop the bleeding before the anoscope is removed. Minor bleeding may also happen for up to two weeks after the biopsy, especially during a bowel movement. Serious bleeding that requires medical attention rarely happens (less than 1% of the time). If you have bleeding that is more than spotting after the procedure, you should call the study clinician.

*Risks to an unborn fetus:* If you become pregnant while taking part in the study, tell the study doctor. There is no known risk of collecting cervical and anal swab specimens or HRA on the pregnancy or unborn fetus. However, HRA evaluations will not be done during pregnancy; only anal Pap and HPV tests will be done.

## What possible benefits can I expect from taking part in this study?

It is possible that you may benefit from this study by being diagnosed for anal or cervical HSIL or pre-cancers. Any treatment will be done outside of the study and may prevent progression to cervical or anal cancers. It is also possible you may receive no benefit from participating. There is a possibility for others infected with HIV and HPV in the future to benefit from this research.

## Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB, FDA, or companies providing the HPV tests

#### What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

| For questions about your rights while in this study, call the | (insert |
|---|---|
| name of center) Institutional Review Board at | (insert telephone number). |
| (Note to Local Investigator: Contact information for patient rep | presentatives or other individuals |
| at a local institution who are not on the IRB or research team | but take calls regarding clinical |
| trial questions can also be listed here.) | |

## What are the costs and payments of taking part in this study?

You will not be asked to pay any costs related to this research. Qiagen Inc., Gen-Probe Inc., and Arbor Vita Corp. are providing the HPV tests at no charge while you take part in this study. However, if you have an abnormal anal Pap or cervical Pap test or biopsy tests, then follow-up care for the abnormal tests are considered standard of care. You and/or your health insurance company will need to pay for the Standard of Care costs.

[Note to local investigator: add language regarding any compensation to subjects for study participation or insert the statement "You will not be paid for taking part in this study."]

## What happens if I am injured because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

# Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor (the AIDS Malignancy Consortium) and its representatives (The EMMES Corporation)
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.

In most cases any health data that is being given out to others is identified by a unique study number and not with your name. Although in some cases it is possible to link your name to the study data, this is not usually done.

# Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Who can answer my questions about the study?

You can talk to your study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor, [name at (###) ###-####].

#### ADDITIONAL STUDIES SECTION:

This section is about optional studies you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will not be added to your medical records and you or your study doctor will not know the results. You will not be billed or receive any payment for taking part in these optional studies. You can still take part in the main study even if you say "no" to any or all of these studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

If you decide you no longer want your samples to be used, you can call the study doctor, (insert name) at (insert telephone number) who will let the researchers know. Then, any sample that remains will no longer be used and related health information will no longer be collected. Samples or related information that have already been given to or used by researchers will not be returned.

Initial your choice for each of the optional studies below.

## 1. Optional future use of samples for other studies by Qiagen

After Qiagen finishes the HPV tests for this study, a portion of your sample will be left over. With your permission, Qiagen would like to keep the leftover sample to run other tests in the future. The future tests are not specified. They may involve cancer screening and prevention, or other research. These studies will not involve genetic testing or growing new cell lines. Qiagen may keep the leftover part of your sample indefinitely. We will not give Qiagen any of your study records or information that links you to your sample. The future testing will be completely anonymous. You will not receive any results of this testing. If you do not agree, Qiagen will not keep any leftover part of your samples.

YES below means that you give permission now. We will not ask again when the specific tests are done. Write your initials below by your choice:

(Initial) YES, I agree to allow Qiagen to keep my leftover samples for future research.

\_\_\_\_\_ (Initial) **NO**, I do not agree to allow Qiagen to keep my leftover study samples.

# 2. Optional AIDS and Cancer Specimen Resource (ACSR) Donation of Leftover Tissue Samples

After all of the tests for this study are finished, there may be unused blood and biopsy tissue left over. We would like your consent to donate your leftover samples to the AIDS and Cancer Specimen Resource (ACSR).

The ACSR is funded by the National Cancer Institute to collect, store, and distribute tissues and

biological fluids from HIV-positive and HIV-negative people to qualified scientists. The ACSR makes these samples available for scientists to do other research studies. This research may be about cancers and pre-cancers associated with HIV disease. The ACSR screens all research plans to be sure that the samples are used to advance scientific research.

Donating your leftover samples to the ACSR will not require any extra tests or procedures. If you do not give your consent, we will destroy your leftover samples at the end of the study.

If you agree to donate leftover samples, we will send them to the ACSR for future use. The ACSR may ask for some medical information from your study records. This information may be useful to researchers who perform studies using your samples. The AMC will not give the ACSR your name or any information that could personally identify you.

We will make every effort to protect your privacy. We will not keep information that links you to your samples after the study is over. You may withdraw your consent to donate your leftover samples at any time during the study. After the study is over, the AMC and the ACSR will not be able to identify your specific samples.

You may contact the research team if you have any questions about donating your leftover samples.

| YES below means that you give permission now. We will not ask again when the specific tests are done. Write your initials below by your choice: |
|---|
| (Initial) YES, I agree to allow ACSR to keep my leftover samples for future research. |
| (Initial) <b>NO</b> , I do not agree to allow ACSR to keep my leftover study samples. |
| This is the end of the section about optional studies. |
| My Signature Agreeing to Take Part in the Main Study |
| I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the main study and any additional studies where I initialed 'yes'. |
| Participant's signature |
| Date of signature |

| sufficient access to i | nformation, incl | uding risks and benefits, to make an informed decision. |
|---|---|---|
| Name of professional | l obtaining conser | nt (print): |
| Signature of person(s | conducting the | informed consent discussion: |
| Date of signature | | |
| In the opinion of th (circle one)? | e Investigator, is | s the participant capable of complying with this protocol |
| YES | NO | |
| Investigator's Name | (print) | Investigator's Signature and Date |

I have fully explained this research study to the subject. In my judgment, there was

## **Attachment 1: AMC Certificate of Confidentiality Statement**

The NIH has given the AMC a Certificate of Confidentiality. The Certificate does not mean that the NIH or the U.S. Government recommend that you take part in this study. This Certificate helps us keep your health information private.

Your records for this study will have information that may identify you. This Certificate lets us turn down legal demands for your study records. We can use the Certificate to turn down demands for records from a U.S. court. The Certificate can be used in any federal, state, or local legal matters. We will use the Certificate to turn down any demands for your study records. The cases where we cannot use the Certificate are explained below.

We cannot use the Certificate to turn down a demand from the U.S. Government for study records. This applies to audits or reviews of the AMC. This also applies to study records that we have to report to the FDA.

The Certificate does not stop you or your family members from sharing your health information. It does not stop you from talking about taking part in this study. You may give written permission for an insurer, employer, or other person to get copies of your study records. If you give permission, we cannot use the Certificate to say no to a request for your study records.